CLINICAL TRIAL: NCT00735761
Title: A Randomized, Double-Blind, Active-Controlled, Subject Initiated Study Comparing ME-609 to Acyclovir Cream for Treatment of Recurrent Herpes Simplex Labialis in Immunocompromised Patients
Brief Title: Study of ME-609 and Acyclovir for Treatment of Herpes Simplex Labialis in Immunocompromised Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Börje Darpö, MD, PhD, Development
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 609-06
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis | interventions — ME 609; Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ME-609 (5% acyclovir and 1% hydrocortisone)
  Interventions: Drug: ME-609
- 2 (Active Comparator): Acyclovir in ME-609 vehicle (5% acyclovir)
  Interventions: Drug: Acyclovir in ME-609 vehicle (5% acyclovir)

INTERVENTIONS:
Drug: ME-609 — Dosage form: Cream Dose and regimen: 5 times daily during 5 days Route of administration: Topical application
  Arms: 1
Drug: Acyclovir in ME-609 vehicle (5% acyclovir) — Dosage form: Cream Dose and regimen: 5 times daily during 5 days Route of administration: Topical application
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the episode duration of a herpes labialis recurrence in immunocompromised patients treated with ME-609 or Acyclovir.

DETAILED DESCRIPTION:
The objective of this study was to evaluate the episode duration of a herpes labialis recurrence, following a 5-day treatment with 5-time daily topical administration of ME-609 or acyclovir cream, in immunocompromised adults, 18 years and older.

This interim report summarizes the results for short-term observations, i.e., during the initial study recurrence. A final study report will be prepared when the long-term follow-up is completed.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent herpes labialis with at least two recurrences during the twelve months prior to the study.
* Stable HIV infection
* CD4+ T-cell count 100 to 500/mm3

Exclusion Criteria:

* Systemic treatment with other antiviral agent or corticosteroids within two weeks prior to and during the treatment period, except for antiretroviral treatment in HIV subjects
* Topical treatment with other antiviral agent or corticosteroids within in or around the oral area within two weeks prior to study drug administration
* Significant skin condition that occur in the area typically affected by herpes recurrences
* Nursing or pregnancy
* Concurrent cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2006-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary variable was episode duration, measured from the start of treatment until loss of hard crust for an ulcerative recurrence and from the start of treatment to time of no signs or symptoms for a non-ulcerative recurrence (Investigator-assessed). | from start of treatment until loss of hard crust

SECONDARY OUTCOMES:
The secondary variable was the time to next recurrence measured from the start of the study recurrence until the start of the next recurrence. | Start of recurrence until start of next recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Anders Sönnerborg, MD PhD Prof., Principal Investigator — Clinical Virology, F68, Karolinska University Hospital, Huddinge, 141 86 Stockholm, Sweden